CLINICAL TRIAL: NCT01647880
Title: Phase II/III Study to Investigate the Effects of Fingolimod Versus Interferon Beta-1b on Visual Recovery After Optic Neuritis
Brief Title: MOdification of VIsual Outcomes After Optic Neuritis in CIS or MS by Gilenya (MOVING Study)
Acronym: MOVING
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: delayed recruitment
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, Friedemann Paul, Sponsor Deputy, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOVING
Record Dates: First submitted 2012-07-23; First posted 2012-07-24 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fingolimod (Gilenya®) (Experimental): 0,5 mg once a day in the morning, oral
  Interventions: Drug: Verum arm receiving Gilenya®
- Interferon beta-1b (Extavia®) (Active Comparator): every second day, s.c.
  Interventions: Drug: Active Comparator receiving Extavia®

INTERVENTIONS:
Drug: Verum arm receiving Gilenya®
  Arms: Fingolimod (Gilenya®)
Drug: Active Comparator receiving Extavia®
  Arms: Interferon beta-1b (Extavia®)

SUMMARY:
In the MOVING study should be examined, whether early therapeutic intervention with fingolimod (Gilenya ®) after optic neuritis(ON) has a favorable visual outcome as a comparative therapie with Interferon beta-1b (Extavia®), as measured by multifocal visual evoked potentials (mVEP) after 6 month compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing-remitting multiple sclerosis (RRMS)
* ability to consent and a written approval
* First acute ON attack to the fit eye within 30 days before screening
* Age 18 - 55 years at screening
* EDSS ≤ 6.0
* No MS Attack except for ON in the last 30 days before screening
* No immunomodulatory therapy for at least three Months (before randomization), or
* strong immunomodulatory therapy with interferon beta or glatiramer acetate for at least 6 months
* visus in the affected eye at least 0.1
* latency of Conventional VEP in the affected eye

  * = 115 ms or difference> = 15 ms to the opposite side at a Study at least 4 but no more than 6 weeks after Onset of clinical symptoms
* At least 2 T2 lesions typical of MS in a previous MRI

Exclusion Criteria:

* other MS course than RRMS
* any condition which could interfere or prevent the MRI study or other investigations
* known allergy or intolerance, or other contraindication against Gd-DTPA
* Patients with known contraindications to treatment with fingolimod (Gilenya ®) or interferon beta-1b Extavia ®
* Competing diseases which could affect visual functions such as diabetic, retinopathy, glaucoma, retinal detachment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Efficacy parameters
  Decrease of latency of mVEP of the affected eye after 6 months treatment with Gilenya® vs. Extavia® compared to baseline

SECONDARY OUTCOMES:
Efficacy parameters
  Decrease in the latency of the mVEP from the affected eye at the time points 1, 3 and 12 months in comparison to baseline. Retinal nerve fiber layer thickness and macular volume in OCT, visual contrast sensitivity, visual field, Color vision, visual quality of life, in CMRT lesion load in cMRT , neurotrophic factors and axonal damage markers (neurofilament) and neurotrophins (for example, BDNF) in the serum

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Hoffmann, PD Dr. med., Study Director — Charite- NeuroCure
Locations (2):
- Germany (2):
  - Charité-Universitätsmedizin Berlin, Berlin
  - Sankt Josefs Krankenhaus Potsdam Neurologie, Potsdam

REFERENCES:
- [Derived] Albert C, Mikolajczak J, Liekfeld A, Piper SK, Scheel M, Zimmermann HG, Nowak C, Dorr J, Bellmann-Strobl J, Chien C, Brandt AU, Paul F, Hoffmann O. Fingolimod after a first unilateral episode of acute optic neuritis (MOVING) - preliminary results from a randomized, rater-blind, active-controlled, phase 2 trial. BMC Neurol. 2020 Mar 3;20(1):75. doi: 10.1186/s12883-020-01645-z. PMID 32126977